CLINICAL TRIAL: NCT00734266
Title: Changes in Leukotrienes During Cardiac Surgery in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Marcos Vidal Melo, Associate Professor of Anesthesia, Massachusetts General Hospital
Other Study IDs: 2007-P-000164/7
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-03

CONDITIONS: Lung Dysfunction; Inflammatory Response During Cardiac Surgery
Keywords: COPD; CPB; Leukotrienes
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1 Control: Patients with and without chronic obstructive pulmonary disease diagnosed before scheduling for cardiac surgery.
- 2 COPD: Patients with and without chronic obstructive pulmonary disease diagnosed before scheduling for cardiac surgery.

SUMMARY:
The hypotheses of this study are that:

* Production and release of inflammatory substances called leukotrienes are increased during heart surgery with use of a heart-lung machine in humans;
* The increase in these leukotrienes levels after heart surgery is higher in patients with bronchitis and/or emphysema than in patients without previous history of lung disease;
* Levels of leukotrienes are directly correlated with worsening of lung function during and after heart surgery.

DETAILED DESCRIPTION:
In this project, we will test the hypothesis that cys-leukotrienes are released and correlated with the impairment of the lung function after cardiac surgery in patients with COPD. If such hypothesis is substantiated in the study, it would allow us to propose the use of leukotriene inhibitors in the peri-operative period to improve pulmonary function and to decrease complications after cardiac surgery in COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients schedules to undergo cardiac surgery with use of CPB.

Exclusion Criteria:

* inability to provide consent;
* previous diagnosis of asthma;
* acute pre-operative respiratory failure;
* emergency surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients schedules to undergo cardiac surgery with use of CPB.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2007-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
urine cysteinyl leukotriene | intra-operative

CONTACTS AND LOCATIONS:
Overall Officials: Marcos F Vidal Melo, MD, Principal Investigator — Massachusetts General Hospital